CLINICAL TRIAL: NCT07125131
Title: Effects of "Gamification-Enhanced Problem-Based Learning" on Critical Thinking Disposition, Metacognitive Awareness and Clinical Competence Among Nursing Students in Hong Kong
Brief Title: Gamification-Enhanced Problem-Based Learning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UW 24-673
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Gamification; Nursing Education
Keywords: gamification

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamification-Enhanced Problem-Based Learning (Experimental): Five weekly gamification-enhanced problem-based learning program
  Interventions: Other: Gamification-Enhanced Problem-Based Learning
- Lecture (Other): Conventional teaching (didactic lectures) delivered by PowerPoint presentation
  Interventions: Other: Conventional didactic lecture (usual practice)

INTERVENTIONS:
Other: Gamification-Enhanced Problem-Based Learning — An educational intervention combines principles of problem-based learning (PBL) with game design elements including scores, leaderboards, digital badges, challenges, immersive experiences, feedback and rewards into problem-based learning.
  Arms: Gamification-Enhanced Problem-Based Learning
Other: Conventional didactic lecture (usual practice) — A didactic teaching approach in which course content is delivered to nursing students primarily through PowerPoint presentation by lecturer.
  Arms: Lecture

SUMMARY:
The goal of this randomized controlled trial is to compare the effects of "Gamification-Enhanced Problem-Based Learning" and a lecturing approach on critical thinking disposition, metacognitive awareness and clinical competence among nursing students of enrolled nurse in higher diploma education in Hong Kong. The main questions it aims to answer are:

1. What is the level of critical thinking disposition, metacognitive awareness and clinical competence of nursing students of enrolled nurse in higher diploma education in Hong Kong?
2. What is the relationship of clinical competence is related to critical thinking disposition and metacognitive awareness among nursing students of enrolled nurse in higher diploma education in HK?
3. What are the effects of "Gamification-Enhanced Problem-Based Learning" and lecturing approach on critical thinking disposition, metacognitive awareness and clinical competence among nursing students of enrolled nurse in higher diploma education in Hong Kong?

Participants will receive five sessions of "Gamification-Enhanced Problem-Based Learning" for five weeks.

DETAILED DESCRIPTION:
A "Gamification-Enhanced Problem-Based Learning" will be provided to the nursing students in a face-to-face format in a local nursing school over five weeks. The duration of each session is 90 mins. The program will take place outside regular class teaching hours and does not contribute to any academic grade points.

The problem-based learning was gamified by designing five levels of authentic clinical cases with increasing difficulties were developed for the program to reflect the clinical situations in real life. Pre-reading materials, which are relevant to the clinical cases, will be given to the participants through an online learning platform one week before each session to support students' learning. The participants, randomly allocated in a group of 4-6 individuals, will work collaboratively to solve the clinical case presented. The process of problem-based learning will be facilitated by a nurse educator. Participants will be allowed to use digital devices e.g. iPad for online resources. Within the one-hour time limit, participants have to put their thinking into action through role-play in the nursing laboratory. The participants will randomly pick their roles e.g. patient's daughter, nurse-in-charge, wound care nurse, observer etc. A patient simulator will be act as a patient to ensure consistency for each group. Relevant medical equipment will be provided to further enhance the immersive experiences. A 20 mins debriefing session will be conducted to consolidate their learning and provide feedback. After completion of a case, a digital badge will be issued to the participants through the online learning platform.

The time used to solve each case will be recorded and converted into score, displaying in leaderboard each week in the online learning platform. The fastest group will be the winner of the program and a certificate of champion will be issued. For those participants who completed all cases will also be awarded a certificate of completion.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or above;
* year 2 nursing students from full-time program;
* education level post-secondary school or above;
* consent given to participate voluntarily in this study;
* participants who could read and write Chinese.

Exclusion Criteria:

* healthcare working experience prior to enrollment into the undergraduate nursing program;
* repeater.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Critical thinking disposition | Baseline, immediate after the intervention at week 5, and one month after the completion of intervention at week 9
  The critical thinking disposition will be measured by The California Critical Thinking Disposition Inventory (CCTDI). It is a 75-item scale tool with seven subscales: "Truth-seeking", "Open-mindedness", "Analyticity", "Systematicity", "Confidence in reasoning", "Inquisitiveness" and "Maturity of judgment".

SECONDARY OUTCOMES:
Metacognitive awareness | Baseline, immediate after the intervention at week 5, and one month after the completion of intervention at week 9
  Metacognitive awareness will be measured by Metacognitive Awareness Inventory (MAI). It is a 52-item Likert scale tool with two subscales: "knowledge of cognition" (17 items) and "regulation of cognition" (35 items).
Clinical competence | Baseline, immediate after the intervention at week 5, and one month after the completion of intervention at week 9
  The clinical competence will be measured by the Nurse Professional Competence Scale Short Form (NPC Scale-SF). It is a 35-item Likert scale tool with six subscales: "Nursing Care", "Value-based Nursing Care", "Medical and Technical Care", "Care Pedagogics", "Documentation and Administration of Nursing Care", and "Development, Leadership, and Organization of Nursing Care".

CONTACTS AND LOCATIONS:
Overall Officials: Wing Yee Tun, MNurs, Principal Investigator — Hong Kong Sanatorium & Hospital
Locations (1):
- School of Nursing, Hong Kong Sanatorium & Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No